CLINICAL TRIAL: NCT01516008
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Tapentadol Immediate-Release Formulation in the Treatment of Acute Pain From Bunionectomy; Bridging Study for Korea
Brief Title: A Study of Tapentadol Immediate-Release in the Treatment of Patients With Acute Pain From Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100459; R331333PAI3030 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-03

CONDITIONS: Hallux Valgus
Keywords: Hallux Valgus; Bunionectomy; Bunion; Acute pain; Tapentadol; Tapentadol IR
MeSH Terms: conditions — Hallux Valgus; Bunion; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tapentadol IR 50 mg (Experimental)
  Interventions: Drug: Tapentadol IR 50 mg
- Tapentadol IR 75 mg (Experimental)
  Interventions: Drug: Tapentadol IR 75 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapentadol IR 50 mg — Type= exact number, unit= mg, number= 50, form= tablet, route= oral use. Tapentadol IR will be administered as a single oral dose once every 4 to 6 hours (patients may take their next dose as early as 4 hours, but no later than 6 hours, after the previous dose), for a period of 72 hours.
  Arms: Tapentadol IR 50 mg
Drug: Tapentadol IR 75 mg — Type= exact number, unit= mg, number= 75, form= tablet, route= oral use. Tapentadol IR will be administered as a single oral dose once every 4 to 6 hours (patients may take their next dose as early as 4 hours, but no later than 6 hours, after the previous dose), for a period of 72 hours.
  Arms: Tapentadol IR 75 mg
Drug: Placebo — Form= tablet, route= oral use. Placebo tablets will be administered as a single oral dose every 4 to 6 hours, for a period of 72 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of at least 1 dose of tapentadol IR 50 mg and/or 75 mg versus placebo using the sum of pain intensity difference at 48 hours (SPID48) to measure analgesic effect in Korean patients with acute pain following bunionectomy.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance like flipping a coin), double-blind (neither physician nor patient knows the name of the assigned drug), placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of tapentadol immediate-release (IR) 50 mg and 75 mg in patients who are undergoing bunionectomy (a surgical procedure to remove a bunion). This study was designed to be a similar study to the pivotal global study of PAI-3003/KF32 in order to bridge the results from the global studies and to show similarity in effect of tapentadol between Korean and Caucasian population which will allow extrapolation of the foreign clinical data of tapentadol into Korea. The study will be divided into screening period, surgical period, qualification period, and a double-blind treatment period. The study length, including the screening period, will be up to a maximum duration of 32 days. Eligible patients will be randomly assigned to 1 of 3 treatment groups (tapentadol IR 50 mg, tapentadol IR 75 mg or placebo) in a 1:1:1 ratio. Efficacy and safety assessments will be performed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing primary unilateral first metatarsal bunionectomy that includes a distal Chevron osteotomy only with or without the Akin procedure
* Healthy or medically stable on the basis of clinical laboratory tests performed at screening. If results are outside the normal reference ranges, the patient may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study
* Women must be postmenopausal, surgically sterile, abstinent, or practicing or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study. Women of childbearing potential must have a negative serum β human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test before surgery
* If a male and sexually active, agrees to use an approved method of birth control to prevent pregnancy in his female partner and not to donate sperm from the day of first study drug intake until 3 months after the day of last study drug intake. To qualify for entry into the double-blind treatment period, the following criteria must be met:
* Qualifying baseline pain intensity (PI) must be rated as greater than or equal to 4 on an 11-point (0 to10) PI numerical rating scale (NRS), recorded within 30 minutes before randomization
* Qualifying PI must occur no earlier than 10 hours after the first surgical incision
* Qualifying baseline PI must occur within 9 hours after termination of the systemic analgesia during the postoperative surgical period

Exclusion Criteria:

* History of seizure disorder or epilepsy suggested by the presence of mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening, and/or severe traumatic brain injury, episode(s) of unconsciousness of more than 24 hours duration, or posttraumatic amnesia of more than 24 hours duration within 15 years of screening
* History of malignancy within the past 2 years before the start of the study
* Evidence of active infections that may spread to other areas of the body or a history of human immunodeficiency virus 1 or 2
* Clinical laboratory values reflecting severe renal insufficiency
* Moderately or severely impaired hepatic function, or patients with abnormal alanine aminotransaminase or aspartate aminotransferase
* Clinical laboratory values outside acceptable limits for surgery in the opinion of the investigator
* A clinically significant disease that in the investigator's opinion may affect efficacy or safety assessments
* Treated with anticonvulsants, monoamine oxidase inhibitors, tricyclic antidepressants, neuroleptics, or serotonin norepinephrine reuptake inhibitor within 2 weeks before randomization
* Systemic steroid therapy, excluding inhalers or topical steroids, within the 4 weeks before screening
* Women who plan to become pregnant during the study, or who are breast feeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- South Korea (7):
  - Busan
  - Chungcheongbuk-Do
  - Gwangju
  - Gyeonggi-do
  - Pusan
  - Seoul
  - Ulsan

REFERENCES:
- [Derived] Lee YK, Ko JS, Rhim HY, Lee EJ, Karcher K, Li H, Shapiro D, Lee HS. Acute postoperative pain relief with immediate-release tapentadol: randomized, double-blind, placebo-controlled study conducted in South Korea. Curr Med Res Opin. 2014 Dec;30(12):2561-70. doi: 10.1185/03007995.2014.954665. Epub 2014 Aug 27. PMID 25133962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 11 January 2012 to 2 February 2013. Participants were recruited at 17 study centers in Korea.
Pre-assignment Details: 353 participants were randomly allocated to the 3 treatment arms. 352 participants received at least 1 dose of the study drug and were included in the intent-to-treat (ITT) analysis set.
Groups:
- Placebo: Each participant received matching placebo once every 4 to 6 hours for 3 days
- Tapentadol IR 50 mg: Each participant received 50 mg of Tapentadol immediate release (IR) once every 4 to 6 hours for 3 days
- Tapentadol IR 75 mg: Each participant received 75 mg of Tapentadol immediate release (IR) once every 4 to 6 hours for 3 days
Period: Overall Study
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Started | 114 | 121 | 117
Completed | 69 | 105 | 99
Not Completed | 45 | 16 | 18
Not completed — Adverse Event | 0 | 2 | 7
Not completed — Lack of Efficacy | 44 | 14 | 10
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Reason not specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg | Total
Number analyzed (Participants) | 114 | 121 | 117 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.62) | 51.8 (11.9) | 50.7 (13.45) | 51.3 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 114 | 108 | 331
  Male | 5 | 7 | 9 | 21
Region of Enrollment [Number; unit: participants]
  Korea, Republic Of | 114 | 121 | 117 | 352
Age Customized [Number; unit: participants]
  <65 years | 103 | 105 | 99 | 307
  >=65 years | 11 | 16 | 18 | 45

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Differences (SPID) Over 48 Hours
Description: Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted Sum of PID scores over 48 hours. Total score ranges from -480 (worst) to 480 (best) for SPID48. A higher value of SPID indicates greater pain relief.
Time Frame: 48 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomized participants with at least 1 dose of study medication. Last-observation-carried-forward imputation method used for missing values.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Scores on a scale | 65.3 (121.04) | 131.7 (107.19) | 154.5 (124.03)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value adjusted for multiple treatment group comparisons using the Hochberg method; ANCOVA model with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 76.35, 95% CI 2-sided [51.0 to 101.7] — Difference is SPID48 in tapentadol IR group minus SPID48 in placebo group
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is adjusted for multiple treatment group comparisons using the Hochberg method; ANCOVA model with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 90.60, 95% CI 2-sided [65.1 to 116.1] — Difference is SPID48 in tapentadol IR group minus SPID48 in placebo group

2. Secondary Outcome: Time to First Rescue Medication Use
Description: Rescue medication was defined as any analgesic medication used for participants discontinued due to lack of efficacy (including those started at time of discontinuation) or analgesic medication used during the double-blind period for completed participants.
Time Frame: Up to 48 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomized participants with at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Hours | NA [6.7 to NA] — The median time to the first rescue medication could not be calculated for the treatment group because less than 50 percent of participants (38.6 percent) used rescue medication. | NA [NA to NA] — The median time to the first rescue medication could not be calculated for the treatment group because less than 50 percent of participants (14.0 percent) used rescue medication. | NA [NA to NA] — The median time to the first rescue medication could not be calculated for the treatment group because less than 50 percent of participants (9.4 percent) used rescue medication.
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; Test type: Superiority or Other; p < 0.001, Log Rank — P-value adjusted for multiple treatment group comparisons using the Hochberg method; Stratified by center
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; Test type: Superiority or Other; p < 0.001, Log Rank — P-value adjusted for multiple treatment group comparisons using the Hochberg method; Stratified by center

3. Secondary Outcome: Percent Reduction in Pain Intensity From Baseline at 12, 24, 48, and 72 Hours
Description: Pain intensity was assessed on a 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Participants with no assessment at the given time point, who used an analgesic medication prior to the time point, or who had worse pain intensity at the time point compared to baseline were assigned a percent reduction of 0 percent.
Time Frame: Baseline (Day 1) and 12, 24, 48, and 72 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomized participants with at least 1 dose of study medication.
Measure: Median (Inter-Quartile Range); unit: Percentage Reduction
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Percentage Reduction
  12 hours | 0.0 [0.0 to 30.0] | 28.6 [0.0 to 50.0] | 28.6 [12.5 to 60.0]
  24 hours | 20.0 [0.0 to 50.0] | 44.4 [22.2 to 60.0] | 50.0 [25.0 to 71.4]
  48 hours | 41.4 [0.0 to 71.4] | 66.7 [42.9 to 80.0] | 70.0 [40 to 83.3]
  72 hours | 60.0 [0 to 85.7] | 77.8 [57.1 to 90.0] | 80.0 [50.0 to 90.0]
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; 12 hours; Test type: Superiority or Other; p < 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; 12 hours; Test type: Superiority or Other; p < 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 3: Comparison: Placebo vs Tapentadol IR 50 mg; 24 hours; Test type: Superiority or Other; p = 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 4: Comparison: Placebo vs Tapentadol IR 75 mg; 24 hours; Test type: Superiority or Other; p < 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 5: Comparison: Placebo vs Tapentadol IR 50 mg; 48 hours; Test type: Superiority or Other; p < 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 6: Comparison: Placebo vs Tapentadol IR 75 mg; 48 hours; Test type: Superiority or Other; p < 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 7: Comparison: Placebo vs Tapentadol IR 50 mg; 72 hours; Test type: Superiority or Other; p = 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction
Statistical Analysis 8: Comparison: Placebo vs Tapentadol IR 75 mg; 72 hours; Test type: Superiority or Other; p < 0.001, Log Rank; Between-group comparison of cumulative distributions of percent reduction

4. Secondary Outcome: Response Rate for 30 Percent or Greater Reduction in Pain Intensity at 12, 24, 48, and 72 Hours
Description: Response rate was defined as the percentage of participants with a 30 percent or greater reduction in pain intensity from baseline to 12, 24, 48, and 72 hours. Pain intensity was assessed on a 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Participants with no assessment at the given time point, who used an analgesic medication prior to the time point, or who had worse pain intensity at the time point compared to baseline were assigned a percent reduction of 0 percent.
Time Frame: 12, 24, 48, and 72 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomized participants with at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Percentage of participants
  12 hours | 27.2 | 47.9 | 49.6
  24 hours | 39.5 | 68.6 | 70.9
  48 hours | 53.5 | 79.3 | 76.9
  72 hours | 57.9 | 81.8 | 80.3
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; 12 hours; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; 12 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 3: Comparison: Placebo vs Tapentadol IR 50 mg; 24 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 4: Comparison: Placebo vs Tapentadol IR 75 mg; 24 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 5: Comparison: Placebo vs Tapentadol IR 50 mg; 48 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 6: Comparison: Placebo vs Tapentadol IR 75 mg; 48 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 7: Comparison: Placebo vs Tapentadol IR 50 mg; 72 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 8: Comparison: Placebo vs Tapentadol IR 75 mg; 72 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center

5. Secondary Outcome: Response Rate for 50 Percent or Greater Reduction in Pain Intensity at 12, 24, 48, and 72 Hours
Description: Response rate was defined as the percentage of participants with a 50 percent or greater reduction in pain intensity from baseline to 12, 24, 48, and 72 hours. Pain intensity was assessed on a 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. Participants with no assessment at the given time point, who used an analgesic medication prior to the time point, or who had worse pain intensity at the time point compared to baseline were assigned a percent reduction of 0 percent.
Time Frame: 12, 24, 48, and 72 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomized participants with at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Percentage of participants
  12 hours | 11.4 | 28.9 | 32.5
  24 hours | 31.6 | 46.3 | 54.7
  48 hours | 48.2 | 71.1 | 70.1
  72 hours | 56.1 | 79.3 | 76.9
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; 12 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; 12 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 3: Comparison: Placebo vs Tapentadol IR 50 mg; 24 hours; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 4: Comparison: Placebo vs Tapentadol IR 75 mg; 24 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 5: Comparison: Placebo vs Tapentadol IR 50 mg; 48 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 6: Comparison: Placebo vs Tapentadol IR 75 mg; 48 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 7: Comparison: Placebo vs Tapentadol IR 50 mg; 72 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 8: Comparison: Placebo vs Tapentadol IR 75 mg; 72 hours; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center

6. Secondary Outcome: Sum of Pain Intensity Differences (SPID) Over 12, 24, and 72 Hours
Description: Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. SPID was calculated as the time-weighted Sum of PID scores over 12, 24, and 72 hours. Total score ranges from -120 (worst) to 120 (best) for SPID12, -240 (worst) to 240 (best) for SPID24, -720 (worst) to 720 (best) for SPID72. A higher value of SPID indicates greater pain relief.
Time Frame: 12, 24, and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Scores on a scale
  12 hours | 5.7 (23.59) | 20.4 (22.29) | 24.6 (28.18)
  24 hours | 17.7 (51.88) | 48.1 (47.92) | 60.1 (58.56)
  72 hours | 127.9 (198.61) | 234.5 (170.84) | 264.1 (192.70)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; 12 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 16.52, 95% CI 2-sided [11.1 to 22.0] — Difference is SPID12 in tapentadol IR group minus SPID12 in placebo group
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; 12 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 19.11, 95% CI 2-sided [13.6 to 24.6] — Difference is SPID12 in tapentadol IR group minus SPID12 in placebo group
Statistical Analysis 3: Comparison: Placebo vs Tapentadol IR 50 mg; 24 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 34.71, 95% CI 2-sided [23.2 to 46.2] — Difference is SPID24 in tapentadol IR group minus SPID24 in placebo group
Statistical Analysis 4: Comparison: Placebo vs Tapentadol IR 75 mg; 24 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 43.04, 95% CI 2-sided [31.5 to 54.6] — Difference is SPID24 in tapentadol IR group minus SPID24 in placebo group
Statistical Analysis 5: Comparison: Placebo vs Tapentadol IR 50 mg; 72 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 122.32, 95% CI 2-sided [81.8 to 162.9] — Difference is SPID72 in tapentadol IR group minus SPID72 in placebo group
Statistical Analysis 6: Comparison: Placebo vs Tapentadol IR 75 mg; 72 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 138.57, 95% CI [97.8 to 179.4] — Difference is SPID72 in tapentadol IR group minus SPID72 in placebo group

7. Secondary Outcome: Total Pain Relief (TOTPAR) Over 12, 24, 48, and 72 Hours
Description: Participants rated pain relief rated on 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Total Pain Relief (TOTPAR) was calculated as the time-weighted sum of pain relief scores up to Hour 12, 24, 48, and 72 hours. Total score ranges from 0 (worst) to 48 (best) for TOTPAR12, 0 (worst) to 96 (best) for TOTPAR24, 0 (worst) to 192 (best) for TOTPAR48, and 0 (worst) to 288 (best) for TOTPAR72. A higher value of TOTPAR indicated greater pain relief.
Time Frame: 12, 24, 48, and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Scores on a scale
  12 hours | 7.8 (7.21) | 15.0 (8.94) | 15.1 (9.99)
  24 hours | 19.4 (16.91) | 34.5 (19.04) | 35.1 (19.50)
  48 hours | 53.8 (44.60) | 88.4 (40.24) | 87.6 (41.34)
  72 hours | 94.7 (76.12) | 151.3 (64.14) | 148.5 (65.29)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; 12 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 7.15, 95% CI 2-sided [5.0 to 9.3] — Difference is TOTPAR12 in tapentadol IR group minus TOTPAR12 in placebo group
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; 12 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 7.13, 95% CI 2-sided [4.9 to 9.3] — Difference is TOTPAR12 in tapentadol IR group minus TOTPAR12 in placebo group
Statistical Analysis 3: Comparison: Placebo vs Tapentadol IR 50 mg; 24 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 15.21, 95% CI 2-sided [10.6 to 19.8] — Difference is TOTPAR24 in tapentadol IR group minus TOTPAR24 in placebo group
Statistical Analysis 4: Comparison: Placebo vs Tapentadol IR 75 mg; 24 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 15.54, 95% CI 2-sided [10.9 to 20.2] — Difference is TOTPAR24 in tapentadol IR group minus TOTPAR24 in placebo group
Statistical Analysis 5: Comparison: Placebo vs Tapentadol IR 50 mg; 48 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 34.76, 95% CI 2-sided [24.3 to 45.3] — Difference is TOTPAR48 in tapentadol IR group minus TOTPAR48 in placebo group
Statistical Analysis 6: Comparison: Placebo vs Tapentadol IR 75 mg; 48 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 33.60, 95% CI 2-sided [23.0 to 44.2] — Difference is TOTPAR48 in tapentadol IR group minus TOTPAR48 in placebo group
Statistical Analysis 7: Comparison: Placebo vs Tapentadol IR 50 mg; 72 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 56.59, 95% CI 2-sided [39.4 to 73.8] — Difference is TOTPAR72 in tapentadol IR group minus TOTPAR72 in placebo group
Statistical Analysis 8: Comparison: Placebo vs Tapentadol IR 75 mg; 72 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA including treatment group and center as factors and baseline pain intenstidy as covariate; Mean Difference (Net) = 53.48, 95% CI 2-sided [36.2 to 70.8] — Difference is TOTPAR72 in tapentadol IR group minus TOTPAR72 in placebo group

8. Secondary Outcome: Sum of Pain Relief and Pain Intensity Differences (SPRID) Over 12, 24, 48, and 72 Hours
Description: Participants rated pain relief rated on 5-point categorical scale of 0-4 (0=none, 1=A little, 2=Some, 3=A lot, 4=Complete). Pain Intensity (PI) was assessed on an 11-point numerical rating scale from 0=no pain to 10=pain as bad as you can imagine. PID was the difference between baseline PI (prior to the first dose) and current PI at assessment. PRID is the sum of pain relief and PID at the same assessment time. SPRID was calculated as the time-weighted Sum of PRID scores over 12, 24, 48, and 72 hours. Total score ranges from -120 (worst) to 168 (best) for SPRID12, -240 (worst) to 336 (best) for SPRID24, -480 (worst) to 672 (best) for SPRID48, and -720 (worst) to 1008 (best) for SPRID72. A higher value of SPRID indicates greater pain relief.
Time Frame: 12, 24, 48, and 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Scores on a scale
  12 hours | 13.6 (29.13) | 35.4 (28.74) | 39.7 (36.18)
  24 hours | 37.1 (65.27) | 82.6 (61.99) | 95.2 (74.14)
  48 hours | 119.1 (159.28) | 220.2 (137.54) | 242.1 (157.04)
  72 hours | 222.6 (265.92) | 385.7 (220.15) | 412.6 (244.92)
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; 12 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 23.66, 95% CI 2-sided [16.4 to 30.9] — Difference is SPRID12 in the tapentadol IR group minus SPRID12 in the placebo group
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; 12 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 26.24, 95% CI 2-sided [18.9 to 33.6] — Difference is SPRID12 in the tapentadol IR group minus SPRID12 in the placebo group
Statistical Analysis 3: Comparison: Placebo vs Tapentadol IR 50 mg; 24 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 49.93, 95% CI 2-sided [34.4 to 65.4] — Difference is SPRID24 in the tapentadol IR group minus SPRID24 in the placebo group
Statistical Analysis 4: Comparison: Placebo vs Tapentadol IR 75 mg; 24 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 58.58, 95% CI 2-sided [43.0 to 74.2] — Difference is SPRID24 in the tapentadol IR group minus SPRID24 in the placebo group
Statistical Analysis 5: Comparison: Placebo vs Tapentadol IR 50 mg; 48 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 111.12, 95% CI [76.3 to 145.9] — Difference is SPRID48 in the tapentadol IR group minus SPRID48 in the placebo group
Statistical Analysis 6: Comparison: Placebo vs Tapentadol IR 75 mg; 48 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 124.21, 95% CI 2-sided [89.2 to 159.2] — Difference is SPRID48 in the tapentadol IR group minus SPRID48 in the placebo group
Statistical Analysis 7: Comparison: Placebo vs Tapentadol IR 50 mg; 72 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 178.91, 95% CI 2-sided [122.4 to 235.4] — Difference is SPRID72 in the tapentadol IR group minus SPRID72 in the placebo group
Statistical Analysis 8: Comparison: Placebo vs Tapentadol IR 75 mg; 72 hours; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with treatment group and center as factors and baseline pain intensity as covariate; Mean Difference (Net) = 192.05, 95% CI 2-sided [135.2 to 248.9] — Difference is SPRID72 in the tapentadol IR group minus SPRID72 in the placebo group

9. Secondary Outcome: Patient Global Impression of Change (PGI-C) Score at 72 Hours
Description: The PGI-C is a 7-point scale that requires the patients to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the intervention. The response options are: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse. Higher scores indicate worsening.
Time Frame: Baseline (Day 1) and 72 hours
Population: Intent-to-treat (ITT) analysis set, which included all randomized participants with at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Number analyzed (Participants) | 114 | 121 | 117
Percentage of participants
  Very Much Improved | 28.9 | 44.6 | 46.2
  Much Improved | 23.7 | 36.4 | 37.6
  Minimally Improved | 11.4 | 8.3 | 6.0
  No Change | 21.1 | 5.0 | 6.0
  Minimally Worse | 7.9 | 3.3 | 1.7
  Much Worse | 6.1 | 0.8 | 1.7
  Very Much Worse | 0.9 | 1.7 | 0.9
Statistical Analysis 1: Comparison: Placebo vs Tapentadol IR 50 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center
Statistical Analysis 2: Comparison: Placebo vs Tapentadol IR 75 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Controlling for center

ADVERSE EVENTS:
Time Frame: Up to Day 30
Description: For serious adverse events, events with onset up to 30 days after the last dose were included. For other adverse events, events with onset up to 48 hours after the last dose were included.
Arm/Group | Placebo | Tapentadol IR 50 mg | Tapentadol IR 75 mg
Serious Adverse Events (participants affected / at risk) | 0/114 | 2/121 | 0/117
Other Adverse Events (participants affected / at risk) | 22/114 | 58/121 | 74/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=114) | Tapentadol IR 50 mg (N=121) | Tapentadol IR 75 mg (N=117)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Essential tremor (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=114) | Tapentadol IR 50 mg (N=121) | Tapentadol IR 75 mg (N=117)
Constipation (Gastrointestinal disorders) | 1 | 7 | 8
Nausea (Gastrointestinal disorders) | 8 | 44 | 52
Vomiting (Gastrointestinal disorders) | 4 | 14 | 26
Pyrexia (General disorders) | 11 | 5 | 8
Procedural dizziness (Injury, poisoning and procedural complications) | 3 | 14 | 22
Dizziness postural (Nervous system disorders) | 0 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days